CLINICAL TRIAL: NCT06375252
Title: Evaluation of Central Jugular Vein Catheter Lumen Holder Design and Ergonomic Use
Acronym: CJVClumen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Yasemin Özkan, phd student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: sbughfyaseminozkan1985
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Central Venous Catheterization
Keywords: Design, Equipment; Nursing Research; Central Venous Catheterizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention-control group (Experimental): Participants assigned to the intervention-control group of the study performed activities using the central jugular vein catheter lumen retainer apparatus.
  Interventions: Other: Central Jugular Vein Catheter Lumen Holder Apparatus
- control-intervention group (No Intervention): Participants in the control-intervention group first performed the activities without the central jugular vein catheter lumen retainer apparatus, and then performed the activities with the apparatus.

INTERVENTIONS:
Other: Central Jugular Vein Catheter Lumen Holder Apparatus — Participants will experience the central jugular vein catheter lumen holder apparatus, perform walking, sitting, supine, right and left side lying activities and fill out the evaluation forms prepared by the researcher. They will then experience the same activities without the apparatus.
  Arms: intervention-control group

SUMMARY:
The aim of this study was to evaluate the design and ergonomic use of central jugular vein catheter lumen holder.

DETAILED DESCRIPTION:
Central venous catheterisation is one of the invasive procedures commonly used in the treatment and care of patients in internal and surgical clinics and generally in intensive care units and in the follow-up of patients to be operated. Central venous catheters (CVC) are indispensable diagnostic and therapeutic applications in modern medicine. It is a practical method used in cases where venous vessels cannot be used.

Central venous catheterisation is a cannula inserted into the subclavian, jugular or femoral vein. Nurses are responsible for the care and daily control of central venous catheters inserted by physicians. Central venous catheterisation is widely used by nurses in clinical wards, intensive care units and during surgical procedures for many indications such as monitoring, drug administration and parenteral nutrition. Subclavian vein and jugular vein are most commonly used for this purpose. Many complications such as haemothorax, pneumothorax, malposition, air embolism and infection may develop during CVC applications. The role of the nurse is very important in the determination of CVC complications.

In terms of the individual with a central vein catheter, it constitutes a situation where the individual is worried about a catheter placed in his/her body and needs to be sensitive to the area where it is placed. They should be careful while performing daily life activities with the catheter. The presence of the central jugular vein catheter in the neck area affects the head position, and the sagging of the catheter lumens on the dressing causes skin sensitivity.

Individuals with central jugular vein catheters experience some problems such as discomfort due to sagging of the catheter lumens, inability to move comfortably in head and neck movements and sagging of the catheter lumens. The aim of this study was to develop an innovative design of central jugular vein catheter lumen holder to ensure the position, fixation and comfort efficiency of the central jugular vein catheter and to evaluate its ergonomic use.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual over the age of 18
* Not having had a central jugular vein catheter inserted before for any reason (no experience)
* Being literate
* Voluntarily agreeing to participate in the research
* Being able to carry out daily life activities individually

Exclusion Criteria:

* Leaving work voluntarily
* Limitation in the head and neck area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-19 (Estimated); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
demographic information | 10 minutes
  Contains participant identifying information

SECONDARY OUTCOMES:
comfort effect | 30 minutes
  The participant's comfort level is evaluated with Visual Analog Scale.